CLINICAL TRIAL: NCT02064595
Title: TREATMENT OF EXPOSED FRACTURES OF TIBIA: A COMPARATIVE STUDY BETWEEN BIPLANE EXTERNAL FIXATOR AND LOCKED INTRAMEDULLARY NAIL
Brief Title: Open Tibia Fractures a Comparative Study Between Biplane External Fixator and Locked Intramedullary Nail
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fabio lucas rodrigues (Other)
Responsible Party: Sponsor-Investigator, Fabio lucas rodrigues, Md, Faculdade de Medicina do ABC
Organization: Faculdade de Medicina do ABC (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ortofmabc1
Record Dates: First submitted 2014-02-03; First posted 2014-02-17 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Open tíbia Fracture
Keywords: Tibial fractures.; Fracture fixation.; External fixators.; Intramedullary.; Quality of life.
MeSH Terms: conditions — Tibial Fractures | interventions — External Fixators; Fracture Fixation, Intramedullary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intramedullary nail (Other): Fractures treated with intramedullary reamed nail
  Interventions: Procedure: Intramedullary nail
- External fixator (Active Comparator): Tibial fractures treated with biplanar external fixation
  Interventions: Procedure: External fixator

INTERVENTIONS:
Procedure: External fixator — Treatment with external fixation
  Arms: External fixator
Procedure: Intramedullary nail — Fracture treated with intramedullary nail
  Arms: Intramedullary nail

SUMMARY:
The objective of this research is to prospectively evaluate a group of patients with shaft compound fracture of the tibia, treated with a biplanar external fixator or locked intramedullary reamed nail. The investigators evaluate the quality of life, bone healing and postoperative complications.

DETAILED DESCRIPTION:
68 patients will be followed for a minimum of 12 months and a maximum of 24 months.

As inclusion criterion, the investigators considered those with shaft compound fracture of the tibia (occurring two inches below the knee and two inches above the ankle), that per the classification Gustillo and Anderson were grades I, II, and IIIA, in patients with a mature skeleton.

The presence of extensive skin lesions and soft tissue or arterial injury requiring surgical repair (Grades IIIB and C) in the initial care, other fractures with the exception of the fibula, or the presence of wounds with signs of infection in the period between the accident and definitive surgery, were used as exclusion criteria.

The patients will be treated in two ways, biplanar external fixator (Group I) and locked intramedullary reamed nail in the tibia (Group II), being divided into these groups by simple randomization.

During initial care in the emergency room, antibiotic prophylaxis, cleaning, debridement, and external splinting of the fracture were performed by staff on duty. There was no interference with respect to the type of assembly to be used in the initial care, leaving the doctor on duty free to use the type of external fixators which he is most used to.

Patients remained hospitalized and received first-generation cephalosporin and dressing of the wound daily. In the 4th to the 7th postoperative day after the initial procedure, the patient underwent another surgery to reassemble the biplanar external fixation or to convert to the locked intramedullary reamed nail.

External fixation consists of the biplanar assembly with six Schanz pins of six millimeters. The placement of these follows the sequence: two proximal to the fracture in different planes and two distal similar to the first. The investigators performed reduction and placement of two bars, one medial and one lateral. Assessed by radiography, two more pins were then introduced into the medial rod, ending with the fixation of a tube-to-tube rod at the level of the fracture. For fixation by locked intramedullary reamed nail, the access path of introduction used was through the patellar tendon, with the knee flexed at 100 degrees on a radiotransparent table.

ELIGIBILITY:
Inclusion Criteria:

* the investigators considered those with shaft compound fracture of the tibia (occurring two inches below the knee and two inches above the ankle), that per the classification Gustillo and Anderson were grades I, II, and IIIA, in patients with a mature skeleton.

Exclusion Criteria:

* The presence of extensive skin lesions and soft tissue or arterial injury requiring surgical repair (Grades IIIB and C) in the initial care, other fractures with the exception of the fibula, or the presence of wounds with signs of infection in the period between the accident and definitive surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Bone healing | One year
  bone formation in 3 cortical through the fracture in x ray

SECONDARY OUTCOMES:
Quality of life | 1 year
  SF 36

OTHER OUTCOMES:
Infection | 1 year
  Productive fistula, phlogistics signals